CLINICAL TRIAL: NCT00837499
Title: Comparative Study of Breast Cancers and Their Risk Factors Among Mexican Women in Mexico, Mexican-American and African-American Women in the U.S.
Brief Title: Breast Cancers: Risk Factors Among Mexican Women in Mexico, Mexican-American and African-American Women in the U.S.
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2006-0551; 3P50CA116199-02S1 (NIH)
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: Breast; Breast Cancer; Risk Factors; Mexican Women; Mexican-American Women; African-American Women; Epidemiological; Questionnaire; Survey; Interview
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One-time blood draw (about 3 tablespoons). If blood cannot be drawn or not enough blood can be drawn, a saliva sample will be taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mexican Women from Mexico
  Interventions: Behavioral: Questionnaire
- Mexican-American Women in U.S.
  Interventions: Behavioral: Questionnaire
- African-American Women in U.S.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Interview and survey during visit or by phone, 30 - 40 minutes.
  Other Names: Survey

SUMMARY:
The goal of this epidemiologic research study is to find out if various risk factors and certain markers (substances that help identify the presence of cancer) that help predict increased occurrence and prognosis (outcome of disease) of breast cancer differ among Mexican, Mexican-American, and African-American women.

DETAILED DESCRIPTION:
An epidemiologic study looks at the patterns, causes, and control of disease in groups of people. Researchers want to see if various risk factors (such as decreased and delayed fertility, obesity, and a sedentary [low physical activity] lifestyle) and certain markers that cause breast cancer are different in women in the above groups.

If you have breast cancer and you agree to take part in this study, you will be interviewed by a trained interviewer with a questionnaire at a time convenient for you, either during your visit to MD Anderson or The Rose, or by phone. You will be asked questions about your personal demographics (such as your age and race), environmental exposures, medical history, family history of cancer, and other day-to-day lifestyle factors. It should take about 30-40 minutes to complete the interview. Clinical data about your breast cancer treatment will also be collected from your medical records.

You will also have a one-time blood draw (about 3 tablespoons). If blood cannot be drawn or not enough blood can be drawn, you will have a saliva sample taken where you will be required to spit into a container. If you have already donated blood or a saliva sample in the Mexican-American Cohort Study, a portion of that sample may be used instead of having to collect a new sample. Your blood or saliva sample will be used to look at your DNA (genetic material of cells). The study pathologist will look at possible prognostic markers (substances that predict outcome of disease) from tissue obtained from your surgery.

Neither you nor your regular doctor will receive reports of this research study. The results of this research study will not be placed in your health records. All of your information obtained in this study will be kept confidential either in a password-protected computer or in a locked file cabinet in a secure location.

Your participation will be over in this study when all the data has been collected and analyzed.

This is an investigational study. Up to 1,825 women will take part in this multicenter study. Up to 1125 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All women of Mexican and African descent ages 18 years or older.
2. Diagnosis of invasive breast cancer (histologically confirmed invasive adenocarcinoma, including ductal, lobular, medullary, tubular and mucinous cellular patterns) within the past 24 months.
3. Willing to complete a questionnaire.
4. Consent to tissue acquisition (remaining after surgery or preoperative core needle biopsy).

Exclusion Criteria:

1. Male gender
2. Inadequate tissue obtained for the four main clinical markers (ER, PR, Her-2/neu and Ki67).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Woman, 18 years or older, of Mexican descent (Mexican or Mexican-American) or an African-American woman, and have invasive breast cancer during past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 938 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Categorical Response Variables | 5 years

SECONDARY OUTCOMES:
Expression of a breast tumor phenotype marker (expressed versus not expressed) | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Abenaa M. Brewster, MD, MHS, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (4):
  - Arizona Cancer Center, Tucson, Arizona
  - LBJ Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The Rose Diagnostic Center, Houston, Texas
- Mexico (3):
  - University of Sonora, Hermosillo, Sonora
  - Instituto Tecnologico, Ciudad Obregón
  - University of Guadalajara, Guadalajara

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org